CLINICAL TRIAL: NCT00264459
Title: A Multicentre, Placebo-controlled, Double-blind Study to Evaluate Efficacy and Safety of a Perennial Sublingual Specific Immunotherapy With a Liquid Formulation of an Extract of a Six Grass Pollen-mixture in Patients With Clinically Relevant Grass Pollen Sensitivity.
Brief Title: Safety and Efficacy of a Sublingual Specific Immunotherapy With an Extract of a Six Grass Pollen Mixture
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Al0102st
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Grass Pollen Allergy
Keywords: Sublingual immunotherapy; Rhinoconjunctivitis; Rhinitis; Asthma
MeSH Terms: conditions — Rhinitis; Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo was given the same way as a sublingual preparation.
  Interventions: Other: Comparator
- Liquid formulation of an extract of a 6 grass pollen mixture (Experimental): Sublingual application containing allergen extracts of 6 grass pollen species (Holcus lanatus, Dactylus glomerata, Lolium perenne, Phleum pratense, Poa pratensis, Festuca pratensis) pollen allergen extract.
  The study solution was applied sublingually, kept under the tongue for 3 minutes, and swallowed thereafter. Initial treatment was applied on the first day of treatment with a starting dose of 25% of the maintenance dose. Increasing doses of 50% were applied with the second and 100% with the third dose to give the maximum (=maintenance) dose. This was followed by a daily patient selfadministered treatment with the maintenance dose.
  Interventions: Biological: Grass pollen formulation

INTERVENTIONS:
Biological: Grass pollen formulation — Solution for sublingual application containing allergen extracts of 6 grass pollen species (Holcus lanatus, Dactylus glomerata, Lolium perenne, Phleum pratense, Poa pratensis, Festuca pratensis) pollen allergen extract.
  The study solution was applied sublingually, kept under the tongue for 3 minutes, and swallowed thereafter.
  Other Names: specific immunotherapy
  Arms: Liquid formulation of an extract of a 6 grass pollen mixture
Other: Comparator — Solution for sublingual application containing Placebo. The study solution was applied sublingually, kept under the tongue for 3 minutes, and swallowed thereafter.
  Other Names: Specific Immunotherapy
  Arms: Placebo

SUMMARY:
The trial is performed to asses efficacy and safety of a sublingual extract of a six grass pollen mixture

ELIGIBILITY:
Inclusion Criteria:

Rhinitis, Rhinoconjunctivitis, Positive Rast result to grass pollen, Positive skin prick test to grass pollen, Positive specific provocation to grass pollen,

Exclusion Criteria:

Serious chronic diseases, Other perennial allergies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2003-02; Primary Completion 2008-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Symptom and Medication Score (SMS) | 1.5 years of therapy
  The primary endpoint is the change of the area under the curve (AUC, derived from an analysis period of 42 days) of the daily sum of the Symptom and Medication Score (SMS) from the baseline measurement to the measurement after 1.5 years of therapy.

SECONDARY OUTCOMES:
Visual Rating Scale | 1.5 years
  Patients' Assessment of severity of symptoms at the end of each season on a 10 points visual rating scale (VRS)

CONTACTS AND LOCATIONS:
Overall Officials: Ludger Klimek, M.D., Principal Investigator
Locations (1):
- Allergopharma GmbH & Co. KG, Reinbek, Germany

REFERENCES:
- [Result] Worm M. Efficacy and tolerability of high dose sublingual immunotherapy in patients with rhinoconjunctivitis. Eur Ann Allergy Clin Immunol. 2006 Dec;38(10):355-60. PMID 17274520
- [Result] Pfaar O, Klimek L. Efficacy and safety of specific immunotherapy with a high-dose sublingual grass pollen preparation: a double-blind, placebo-controlled trial. Ann Allergy Asthma Immunol. 2008 Mar;100(3):256-63. doi: 10.1016/s1081-1206(10)60451-6. PMID 18426146
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de